CLINICAL TRIAL: NCT00881348
Title: Dermatological Evaluation of the Photo Irritation and Photo Sensitivity Potential for Dermacyd Infantile (Lactic Acid).
Brief Title: Dermacyd Infantile (Lactic Acid) - Photo Evaluation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04680
Record Dates: First submitted 2009-04-10; First posted 2009-04-15 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Hygiene

ARMS (1):
- Dermacyd infantile (Lactic Acid) (Experimental): 5 weeks treatment
  Interventions: Drug: LACTIC ACID(ND)

INTERVENTIONS:
Drug: LACTIC ACID(ND) — Dermacyd infantile (Lactic Acid)

SUMMARY:
Primary Objective:

To demonstrate the absence of photo irritation and photosensitization potential of the product Dermacyd Infantile (Lactic Acid).

ELIGIBILITY:
Inclusion criteria:

* Phototype Skin I, II, III and IV
* Integral skin test in the region
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion.

Exclusion criteria:

* Use of Anti-inflammatory, immunosuppressant or anti-histaminic drugs
* Lactation or gestation
* Use of Anti-inflammatory drugs 30 days and/or immunosuppressant drugs during 3 months before the selection
* Diseases which can cause immunity decrease, such as HIV, diabetes
* Previous atopy
* History of sensitivity or irritation for topic products
* Active cutaneous diseases which can interfere in the study results
* Use of new drugs and/ or cosmetics during the study
* Cutaneous reactivity
* Previous participation in studies, which had used the product
* Volunteers who have immunodeficiency congenital or acquired.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The photo irritation test and the photosensitivity will be measured using UVA irradiation and evaluated according International Contact Dermatitis Research Group (ICDRG) scale. The sensibility will be evaluated according to the skin type. | During 5 weeks (i.e. treatment period)

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil